CLINICAL TRIAL: NCT02380716
Title: ARISE: Evaluation of the GORE® Ascending Stent Graft in the Treatment of DeBakey Type I/II Aortic Dissection
Status: Active, not recruiting | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBE 14-02
Record Dates: First submitted 2015-02-24; First posted 2015-03-05 (Estimated); Results first posted 2023-02-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Aortic Dissection
Keywords: type A dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (1):
- GORE® Ascending Stent Graft (Experimental): Treatment with the GORE® Ascending Stent Graft
  Interventions: Device: GORE® Ascending Stent Graft

INTERVENTIONS:
Device: GORE® Ascending Stent Graft

SUMMARY:
Assess the feasibility of the treatment of DeBakey Type I/II aortic dissections with the GORE® Ascending Stent Graft

DETAILED DESCRIPTION:
This study is a prospective, multicenter, non-randomized single-arm study to assess the feasibility of the treatment of DeBakey Type I/II aortic dissections with the GORE® Ascending Stent Graft.

ELIGIBILITY:
Inclusion Criteria:

1. DeBakey Type I/II aortic dissection compatible with the treatment requirements of GORE® Ascending Stent Graft, including:

   * Primary entry tear must be in the ascending aorta and ≥2cm distal to the most distal coronary artery ostia
   * Ascending aorta compatible with the GORE® Ascending Stent Graft including landing zone true lumen diameter between 24mm - 42mm and total aortic landing zone diameter ≤ 45 mm
2. Able to undergo CT scan per protocol requirements to perform required case planning prior to endovascular procedure
3. High surgical risk, as determined by the implanting physician
4. Adequate vascular access via transfemoral or retroperitoneal approach
5. An Informed Consent Form signed by Subject or legally authorized representative
6. Able to comply with protocol requirements including follow-up

Exclusion Criteria:

1. Planned aortic valve repair or replacement or coronary artery intervention within 30 days
2. Presence of mechanical heart valve in the aortic position
3. Primary entry tear location in the aortic arch or descending thoracic aorta with retrograde flow into the ascending aorta
4. Aortic insufficiency grade 3+ or 4+
5. Known irreversible neurological injury
6. Known degenerative connective tissue disease, e.g. Marfan's or Ehler-Danlos Syndrome
7. Participation in another drug or medical device study within 1 year of study enrollment
8. Known history of drug abuse
9. Pregnant female at time of informed consent signature
10. Body habitus or other medical condition which prevents adequate visualization of the aorta
11. Systemic infection that could increase the risk of endovascular graft infection
12. Previous thoracic aortic surgery
13. Life expectancy <12 months due to associated non-cardiac co-morbid conditions
14. Subject has known sensitivities or allergies to the device materials
15. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin
16. Patient has known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California- Keck Medicine, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GORE® Ascending Stent Graft: Treatment with the GORE® Ascending Stent Graft
  GORE® Ascending Stent Graft
Period: Overall Study
Arm/Group | GORE® Ascending Stent Graft
Started | 21
Primary Endpoint Analyzed | 19
Completed | 1 (Completed to date (Aug 2022))
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.2 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality at 30 Days Post-procedure
Description: Number of subjects that die of any cause within 30 days post-procedure
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 19
Participants | 3

2. Secondary Outcome: Successful Dissection Treatment (Technical Success)
Description: Number of subjects with technical success defined as successful access to the aorta, successful deployment of the study device components, successful retrieval of the device delivery system, exclusion of the primary entry tear of the aortic dissection, and patency of the side branch device component, if used.
Time Frame: At removal of device deployment system, up to conclusion of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 21
Participants | 17

3. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE) Assessed Through 30 Days, 6 Months, and 12 Months
Description: Assessed by reported adverse events that meet the MACCE criteria and adjudicated by a Clinical Events Committee
Time Frame: 30 days, 6 months, and 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 21
Participants | 9

4. Secondary Outcome: Individual MACCE Components Through 30 Days, 6 Months, and 12 Months
Description: Individual Components include: All Cause Mortality, Myocardial Infarction (MI), and Severe Stroke.
  Assessed by reported adverse events that meet the MACCE criteria and adjudicated by a Clinical Events Committee.
Time Frame: 30 days, 6 months, and 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 21
Participants
  All Cause Mortality - Through 30 Days | 3
  All Cause Mortality - Through 6 Months (183 Days) | 4
  All Cause Mortality - Through 1 Year (365 Days) | 4
  Myocardial Infarction - 30 Days | 0
  Myocardial Infarction - 6 Months (183 Days) | 0
  Myocardial Infarction - One Year (365 Days) | 0
  Severe Stroke - 30 Days | 2
  Severe Stroke - 6 Months (183 Days) | 3
  Severe Stroke - One Year (365 Days) | 3

5. Secondary Outcome: Aorta-related Mortality
Description: Assessed by reported adverse events and adjudicated by a Clinical Events Committee
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 21
Participants | 3

6. Secondary Outcome: Number of Participants With Device Migration Assessed Through 1 Month, 6 Months, and 12 Months
Description: Assessed on CT scans within the defined visits windows
  1 Month: 15-59 days post procedure 6 Month: 60-242 days post procedure 12 Month: 243-546 days post procedure
Time Frame: 30 days, 6 months, and 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 21
Participants
  30 Day Device Migration | 0
  6 Month (183) Device Migration | 0
  1 Year (365 Day) Device Migration | 0

7. Secondary Outcome: Endoleak Assessed Through 1 Month, 6 Months, and 12 Months
Description: Assessed on CT scans within the defined visits windows:
  1 Month: 15-59 days post procedure 6 Month: 60-242 days post procedure 12 Month: 243-546 days post procedure
  Definitions:
  Endoleak Type I (A and B): Endoleak arising at or from the prosthesis attachment site perfusing the treated region of the aorta.
  Endoleak Type IA: Endoleak at proximal aortic prosthesis attachment site. Endoleak Type IB: Endoleak at distal prosthesis attachment site. Endoleak Type II: Endoleak arising from a patent branch vessel of the excluded aorta perfusing the treated aorta, e.g., lumbar or inferior mesenteric branch.
  Endoleak Type III: Endoleak arising from the component junction(s) of the prosthesis or due to a defect in the graft material perfusing the treated region of the aorta.
  Endoleak Type IV: Endoleak arising through the graft fabric perfusing the treated region of the aorta.
  ***Endoleak categorizations have no directionality (i.e., cannot be considered better or worse)**
Time Frame: 30 days, 6 months, and 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® Ascending Stent Graft
Number analyzed (Participants) | 21
Participants
  Any Endoleak - 1 Month | 3
  Any Endoleak - 6 Month | 4
  Any Endoleak - 12 Month | 4
  Type IA Endoleak - 1 Month | 3
  Type IA Endoleak - 6 Month | 3
  Type IA Endoleak - 1 Year | 3
  Type IB Endoleak - 1 Month | 0
  Type IB Endoleak - 6 Month | 0
  Type IB Endoleak - 12 Month | 0
  Type II Endoleak - 1 Month | 0
  Type II Endoleak - 6 Month | 0
  Type II Endoleak - 12 Month | 0
  Type III Endoleak - 1 Month | 1
  Type III Endoleak - 6 Month | 2
  Type III Endoleak - 12 Month | 2
  Type IV Endoleak - 1 Month | 0
  Type IV Endoleak - 6 Month | 0
  Type IV Endoleak - 12 Month | 0

ADVERSE EVENTS:
Time Frame: Through 5 Years or Study Discontinuation/Completion
Arm/Group | GORE® Ascending Stent Graft
All-Cause Mortality (participants affected / at risk) | 6/21
Serious Adverse Events (participants affected / at risk) | 19/21
Other Adverse Events (participants affected / at risk) | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® Ascending Stent Graft (N=21)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 5 (7)
Embolic Stroke (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 3 (3)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (2)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Atrial Fibrilation (Cardiac disorders) | 3 (4)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Aortic Rupture (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Calculus Bladder (Renal and urinary disorders) | 1 (1)
Injury Associated with Device (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Infusion Site Extravasation (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Stent-Graft Endoleak (General disorders) | 3 (5)
Device Placement Issue (Injury, poisoning and procedural complications) | 1 (1)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Weaning Failure (Injury, poisoning and procedural complications) | 1 (1)
Arterial Puncture (Surgical and medical procedures) | 1 (1)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® Ascending Stent Graft (N=21)
Clostridium Difficile Colities (Infections and infestations) | 1 (1)
Pneumonia Aspiration (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Accelerated Hypertension (Vascular disorders) | 1 (1)
Aortic Dissection (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Truncus Coeliacus Thrombosis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 (1)
Adverse Drug Reaction (General disorders) | 1 (1)
Stent-Graft Endoleak (General disorders) | 4 (4)
Device Placement Issue (Injury, poisoning and procedural complications) | 1 (1)
Incision Site Swelling (Injury, poisoning and procedural complications) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT02380716/Prot_SAP_001.pdf